CLINICAL TRIAL: NCT07081438
Title: Taking Psychiatry Online: Developing a Platform to Provide Internet-Delivered Cognitive-Behavior Therapy and Testing It in Obsessive-Compulsive Disorder
Brief Title: iCBT for Adult Obsessive-Compulsive Disorder
Acronym: icbtadultOCD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2023/0643
Record Dates: First submitted 2025-07-10; First posted 2025-07-23 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Obsessive-Compulsive Disorder (OCD)
Keywords: Obsessive-Compulsive Disorder; Cognitive-behavior therapy; icbt; Online treatment; e-health
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Single-Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-delivered Cognitive Behavioral Therapy (iCBT) (Experimental)
  Interventions: Behavioral: icbt

INTERVENTIONS:
Behavioral: icbt — 12-Week Therapist-Based iCBT for OCD (Adapted Version of OCD Net: https://therapistguide.webcbt.se/index.html)

SUMMARY:
The goal of the study is to assess the feasibility, acceptability, and potential effects of therapist-guided internet-delivered cognitive-behavior therapy (iCBT) for adult obsessive-compulsive disorder, using a recently developed digital platform.

DETAILED DESCRIPTION:
Although cognitive-behavior therapy (CBT) is a well-established first-line treatment for many mental disorders, very few patients receive it due to the shortage of trained professionals, the costs of face-to-face therapy, and geographic barriers. Therapist-guided internet-delivered CBT (iCBT) is a potential solution to this problem but is not generally available in our context.

The investigators plan to:

1. Develop a digital platform for the treatment of mental disorders using therapist-guided iCBT;
2. Assess the feasibility, acceptability, and potential effects of therapist-guided iCBT for adult obsessive-compulsive disorder (OCD) using the platform developed in Objective 1.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75
* Internet access
* Principal diagnosis of OCD, based on DSM-5
* Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) Total Severity Score > 16
* Ability to communicate in Spanish
* For participants taking psychotropic medication for OCD: at least eight weeks on stable medication and willingness to stay on the same medication/doses for the 12 weeks of the study

Exclusion Criteria:

* Estimated IQ < 70, as per the Vocabulary subtest of the Wechsler Adults Intelligence Scale for Children (WISC)
* Eight or more previous sessions of CBT for OCD with an experienced therapist during the last 12 months
* Ongoing psychological treatment for OCD
* Diagnosis of organic brain disorder, intellectual disability, autism spectrum disorder, psychosis, bipolar disorder, low-weight anorexia nervosa, or alcohol/substance dependence
* Immediate risk to self or others (e.g., suicidality)
* Inability to communicate in Spanish
* Low motivation to participate (i.e., the patient does not believe the therapy will be helpful at all)
* Insufficient time to work on the treatment (about 30 minutes per day)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility (recruitment and retention rates and therapist burden) | From enrollment to the end of treatment at 12 weeks
  The investigators will assess feasibility by recording recruitment rates, retention rates, and therapist burden (time spent by the therapist sending emails, reviewing materials, etc.).

OTHER OUTCOMES:
Acceptability (Treatment Acceptability/Adherence Scale, TAAS) | Immediately after the intervention
  The TAAS assesses satisfaction with treatment and adherence.
Yale-Brown Obsessive-Compulsive Scale | Baseline and 12 weeks
  The Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) evaluates the severity of obsessive-compulsive disorder symptoms in adults. It is a clinician-rated, 10-item scale, with each item rated from 0 (no symptoms) to 4 (extreme symptoms), resulting in a total score ranging from 0 to 40. The scale also provides separate subtotals for the severity of obsessions and compulsions.
Clinical Global Impression (CGI)-Severity | Baseline and 12 weeks
  The CGI rates the severity of the patient's illness at the time of assessment on a 7-point scale, from 1 = normal to 7 = among the most extremely ill patients.
Beck Depression Inventory | Baseline and 12 weeks
  The BDI assesses the severity of depressive symptoms in adolescents and adults.
Negative Effects Questionnaire (NEQ) | Baseline, mid-intervention and 12-weeks
  The NEQ assesses potential negative side effects of the intervention.
Obsessive-Compulsive Inventory Revised (OCI-R) | Baseline and after 12 weeks
  The OCI-R assesses obsessive-compulsive symptoms experienced over the past month. It is an 18-item self-report questionnaire covering six symptom dimensions: washing, checking, ordering, obsessing, hoarding, and neutralizing. Each item is rated on a 5-point scale (0 = not at all, 4 = extremely), reflecting the distress caused by the symptom during the past month.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Radua, MD, Principal Investigator — Instituto de Investigaciones Biomédicas August Pi i Sunyer (IDIBAPS)

IPD SHARING:
Plan to Share IPD: No